CLINICAL TRIAL: NCT05942209
Title: Diagnostic and Preventive Strategies for Colorectal Anastomotic Leakage in Patients With Gynecologic Tumors
Brief Title: ECO-LEAK Technique: Early Detection of Colorectal Anastomotic Leakage by Transvaginal Ultrasound
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Collaborators: Clinica Universidad de Navarra, Universidad de Navarra (Other); Instituto de Investigación Hospital Universitario La Paz (Other); Hospital Universitario Virgen de la Arrixaca (Other); Hospital Universitario 12 de Octubre (Other); Imperial College London (Other); Kliniken Essen-Mitte (Other); Charite University, Berlin, Germany (Other); Instituto Nacional de Cancerologia, Columbia (Other Government); Hospital Britanico (Other); University of the Republic, Uruguay (Other); Hospital Erasto Gaertner (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-837-1; Victor Lago Leal (Other: La Fe)
Record Dates: First submitted 2023-06-14; First posted 2023-07-12 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-01

CONDITIONS: Gynecologic Cancer; Anastomotic Leak; Cytoreductive Surgery
Keywords: transvaginal ultrasound; enema; anastomotic leakage; Computed Tomography Scan (CT-SCAN)
MeSH Terms: conditions — Anastomotic Leak | interventions — Tomography, X-Ray Computed; Proctoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- ECO-LEAK transvaginal ultrasound: A transvaginal ultrasound is performed with a transrectal enema performed routinely during 4th-6th post-operative day
  Interventions: Diagnostic Test: ECO-LEAK transvaginal ultrasound; Diagnostic Test: ECO-LEAK with CT-Scan or rectoscopy; Diagnostic Test: CT-Scan or rectoscopy
- ECO-LEAK with other diagnostic method (Computed Tomography Scan or rectoscopy): Women with colo-rectal anastomosis with a CT-SCAN (Computed Tomography Scan) or rectoscopy image test performed routinely during 4th-6th post-operative day and a transvaginal ultrasound
  Interventions: Diagnostic Test: ECO-LEAK transvaginal ultrasound; Diagnostic Test: ECO-LEAK with CT-Scan or rectoscopy; Diagnostic Test: CT-Scan or rectoscopy
- CT-SCAN and/or rectoscopy: Women with colo-rectal anastomosis with a CT-SCAN or rectoscopy image test performed routinely during 4th-6th post-operative day
  Interventions: Diagnostic Test: ECO-LEAK transvaginal ultrasound; Diagnostic Test: ECO-LEAK with CT-Scan or rectoscopy; Diagnostic Test: CT-Scan or rectoscopy

INTERVENTIONS:
Diagnostic Test: ECO-LEAK transvaginal ultrasound — After performing the colorectal anastomosis, the patient is monitored postoperatively both clinically and analytically, with serial laboratory tests including PCR and procalcitonin. In the absence of symptoms on the 4th to 5th day an ultrasound - ecoenema is performed. First, the Foley catheter is inserted via the transanal route with instillation of 180cc of serum under ultrasound guidance with a probe in the vagina, using a sagittal and midline cut. In case there is the appearance of free pelvic fluid (previously absent) or an increase in free fluid compared to the baseline examination (fluid present at the beginning of the examination) around the anastomosis/pelvic area, the test will be considered positive.
Diagnostic Test: ECO-LEAK with CT-Scan or rectoscopy — After performing the colorectal anastomosis, the patient is monitored postoperatively both clinically and analytically, with serial laboratory tests including PCR and procalcitonin. In the absence of symptoms on the 4th to 5th day, a CT scan or rectoscopy is performed, along with an ecoenema.
Diagnostic Test: CT-Scan or rectoscopy — After performing the colorectal anastomosis, the patient is monitored postoperatively both clinically and analytically, with serial laboratory tests including PCR and procalcitonin. In the absence of symptoms on the 4th to 5th day, a CT scan or rectoscopy is performed

SUMMARY:
The main hypothesis is that anastomotic leakage can be predicted peri- and postoperatively.To this end, the aim is to establish the accuracy of transvaginal ultrasound with transrectal enema (Ecoenema-TV) for the diagnosis of anastomotic leakage in patients undergoing colorectal anastomosis.

diagnosis of anastomotic leakage in patients undergoing colorectal anastomosis.

DETAILED DESCRIPTION:
Cytoreductive surgery is the cornerstone of advanced ovarian cancer treatment and often requires the performance of a modified posterior pelvic exenteration (MPE) or colorectal resection (CRR), ideally followed by an end-to-end colorectal anastomosis with the goal of achieving optimal cytoreduction. One of the most challenging complications of this procedure is anastomotic leakage (AL) which is considered a life-threatening situation with a reported incidence between 1.24% and 9% in patients with ovarian cancer making any adjuvant postoperative treatment challenging and therefore having a negative impact on the overall prognosis.

In order to diagnose the presence of anastomotic leakage in female patients after colorectal anastomosis we devised this diagnostic test during the postoperative period.

The ECO-LEAK test is performed in the following sequence, after informing the patient and obtaining her consent. The patient is placed in gynaecological position/ lithotomy. Then basal transvaginal ultrasound is performed with the aim of describing the presence or absence of free fluid or other ultrasound findings (sagittal and transverse scan). Simultaneously transanal foley catheter is introduced and filled the balloon of the probe by direct visualization. Then transvaginal ultrasound with enema is performed with insertion of 180cc of serum under ultrasound vision with probe in vagina and sagittal and mid-sagittal cut. If no new free peri-anastomotic/pelvic fluid appears, the test is considered negative. If there is an appearance of pelvic free fluid (previously absent) or an increase in free fluid with respect to the baseline examination (fluid present at the beginning of the examination) peri anastomosis/pelvic, the test is considered positive.

In conclusions, anastomotic leak can occur despite a normal intraoperative anastomosis check-up. Transvaginal ultrasound associated with a transrectal enema (ECO-LEAK) performed during post operative period might represent an useful tool for anastomotic leak diagnosis. A prospective study is needed in order to determine its accuracy

ELIGIBILITY:
Inclusion Criteria:

* Woman sex
* Age between 21-99 years old
* Colorectal resection and anastomosis
* Anastomosis upper from 5 cm from anal verge
* Signed informed consent

Exclusion Criteria:

* No colorectal anastomosis after resection
* Ultralow colorectal anastomosis (< 5 cm)
* Insufficient vaginal cuff for TV-US examination

Ages: 21 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with gynecological cancer with colorectal resection and anastomosis
Sampling Method: Non-Probability Sample
Enrollment: 766 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
To ascertain the sensitivity, specificity , positive predictive value and negative predictive value of the test to diagnose an anastomotic leak after colorectal resection during post-operative period | 24 months
  ECO-LEAK for anastomotic leakage diagnosis in women after colorectal resection and anastomosis

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari i Politecnic La Fe, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bristow RE, del Carmen MG, Kaufman HS, Montz FJ. Radical oophorectomy with primary stapled colorectal anastomosis for resection of locally advanced epithelial ovarian cancer. J Am Coll Surg. 2003 Oct;197(4):565-74. doi: 10.1016/S1072-7515(03)00478-2. PMID 14522325
- [Background] Bartl T, Schwameis R, Stift A, Bachleitner-Hofmann T, Reinthaller A, Grimm C, Polterauer S. Predictive and Prognostic Implication of Bowel Resections During Primary Cytoreductive Surgery in Advanced Epithelial Ovarian Cancer. Int J Gynecol Cancer. 2018 Nov;28(9):1664-1671. doi: 10.1097/IGC.0000000000001369. PMID 30371563
- [Background] Valenti G, Vitagliano A, Morotti M, Giorda G, Sopracordevole F, Sapia F, Lo Presti V, Chiofalo B, Forte S, Lo Presti L, Tozzi R. Risks factors for anastomotic leakage in advanced ovarian cancer: A systematic review and meta-analysis. Eur J Obstet Gynecol Reprod Biol. 2022 Feb;269:3-15. doi: 10.1016/j.ejogrb.2021.12.007. Epub 2021 Dec 13. PMID 34942555
- [Background] Lago V, Fotopoulou C, Chiantera V, Minig L, Gil-Moreno A, Cascales-Campos PA, Jurado M, Tejerizo A, Padilla-Iserte P, Malune ME, Di Donna MC, Marina T, Sanchez-Iglesias JL, Olloqui A, Garcia-Granero A, Matute L, Fornes V, Domingo S. Risk factors for anastomotic leakage after colorectal resection in ovarian cancer surgery: A multi-centre study. Gynecol Oncol. 2019 Jun;153(3):549-554. doi: 10.1016/j.ygyno.2019.03.241. Epub 2019 Apr 3. PMID 30952369
- [Background] Lago V, Segarra-Vidal B, Cappucio S, Angeles MA, Fotopoulou C, Muallem MZ, Manzanedo I, Iglesias JLS, Chacon E, Padilla-Iserte P, Fagotti A, Ferron G, Kluge L, Vargiu V, Del M, Scambia G, Minig L, Tejerizo A, Segovia MG, Cascales-Campos PA; OVA-LEAK Collaborative Group; Hervas D, Domingo S. OVA-LEAK: Prognostic score for colo-rectal anastomotic leakage in patients undergoing ovarian cancer surgery. Gynecol Oncol. 2022 Oct;167(1):22-27. doi: 10.1016/j.ygyno.2022.08.004. Epub 2022 Sep 2. PMID 36058743